CLINICAL TRIAL: NCT04387630
Title: Neoadjuvant Chemotherapy With or Without Metformin in Early Breast Cancer.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of Surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.20.05.834
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Breast Cancer
Keywords: breast cancer; metformin; anti-tumor immunity
MeSH Terms: conditions — Breast Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin group (Experimental): metformin 850 mg once daily increased within 3 weeks to a maximum dose of 2550 mg on three divided daily doses.
  Neoadjuvant cytotoxic chemotherapy as per MDT (multi-disciplinary team) decision. Patients scheduled for AC-T (adriamycin, Cyclophosphamide, paclitaxel) or AC (adriamycin, cyclophosphamide) will be eligible to randomization.
  Interventions: Drug: Metformin
- Placebo group (Placebo Comparator): placebo. Neoadjuvant cytotoxic chemotherapy as per MDT(multi-disciplinary team) decision. Patients scheduled for AC-T (adriamycin, Cyclophosphamide, paclitaxel) or AC (adriamycin, cyclophosphamide) will be eligible to randomization.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin — Oral hypoglycemic drug. Initial dose 500-850 mg/d. incrementally increased to a maximum daily dose of 2550 mg in three divided doses.
  Other Names: Glucophage
  Arms: metformin group
Drug: Placebo oral tablet — Simethicone 60 mg three times daily.
  Arms: Placebo group

SUMMARY:
Metformin is a widely used anti-diabetic drug. Several studies have pointed out a potentially beneficial effect of metformin therapy in diabetic cancer patients. Several studies are investigating the anti-tumor effect of metformin in early breast cancer. However, the enhancing effect of metformin on anti-tumor immunity has only been demonstrated in animal models. This study examines the immune effect of metformin in breast cancer patients treated with preoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven breast carcinoma.
* American Society of Anesthesiology (ASA) score I-II.
* Candidate for neoadjuvant chemotherapy as per hospital's protocol.
* Clinically measurable tumor.
* No evidence of distant metastasis.
* Normal renal and liver functions.
* Non-diabetics.

Exclusion Criteria:

* Pregnant or lactating women.
* Metastatic breast cancer patients.
* Patients with hepatic impairment.
* Patients with renal impairment.
* Diabetics.
* Patients unwilling to participate or withdrawing from the trial.
* Psychological/ mental impairment.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-06-05 (Actual); Primary Completion 2022-06-05 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response rate | at three months from starting therapy.
  Response to preoperative therapy as per ultrasonographic tumor size assessment. A responder will have > 50% decrease in the size of the primary tumor without appearance of new lesions.

OTHER OUTCOMES:
T-cell cytotoxic markers. | procedure
  Percentage of cells staining positive per high power field for the T-cell cytotoxic markers (Granzyme-B, Perforin & CD-8) using immunohistochemistry (IHC).

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hussein, MD, PhD, Principal Investigator — Mansoura University Faculty of Medicine
Locations (1):
- Mansoura University Cancer center, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Eikawa S, Nishida M, Mizukami S, Yamazaki C, Nakayama E, Udono H. Immune-mediated antitumor effect by type 2 diabetes drug, metformin. Proc Natl Acad Sci U S A. 2015 Feb 10;112(6):1809-14. doi: 10.1073/pnas.1417636112. Epub 2015 Jan 26. PMID 25624476
- [Background] Pearce EL, Walsh MC, Cejas PJ, Harms GM, Shen H, Wang LS, Jones RG, Choi Y. Enhancing CD8 T-cell memory by modulating fatty acid metabolism. Nature. 2009 Jul 2;460(7251):103-7. doi: 10.1038/nature08097. Epub 2009 Jun 3. PMID 19494812
- [Background] Coyle C, Cafferty FH, Vale C, Langley RE. Metformin as an adjuvant treatment for cancer: a systematic review and meta-analysis. Ann Oncol. 2016 Dec;27(12):2184-2195. doi: 10.1093/annonc/mdw410. Epub 2016 Sep 28. PMID 27681864